CLINICAL TRIAL: NCT00486122
Title: Evaluation of Continuous Symptom Treatment of ADHD: A Placebo-Controlled Double-Blind Assessment of Morning-Dosed or Evening-Dosed Strattera
Brief Title: Evaluation of Continuous Symptom Treatment of ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7972; B4Z-US-LYCC
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride
Drug: Placebo

SUMMARY:
The purpose of this study is to test the hypothesis that atomoxetine administered orally, once a day, at doses up to 1.4 mg/kg/day for approximately 6 weeks given in the morning is superior to placebo in children with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have ADHD that meets disease diagnostic criteria as defined by DSM-IV-Revised
* Males or females who are at least 6 years old and no more than 12 years old prior to visit 2
* Patients must be able to swallow capsules
* Patients must be of normal intelligence in the judgment of the investigator. Normal intelligence is defined as being without evidence of significant general intellectual deficit and expected to achieve a score of 70 or more if formal IQ testing were administered.
* Laboratory results must show no significant abnormalities (significance is defined as laboratory values requiring acute medical intervention, indicating a serious medical illness, or requiring further medical evaluation in the judgment of the investigator)

Exclusion Criteria:

* Patients who weigh less than 20 kg or greater than 65 kg at study entry (visit 1)
* Patients who have a documented history of bipolar I or bipolar II disorder, or psychosis
* Patients who have documented autism, Asperger's syndrome, or pervasive developmental disorder.
* Other comorbid psychiatric disorders are not excluded provided that the diagnosis of ADHD predates the comorbid disorder, and that the ADHD symptoms are the primary source of impairment for the patient
* Patients taking any antipsychotic medication during the 4 weeks prior to visit 1 are not eligible.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 282 (Actual)
Dates: Start 2003-09; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that atomoxetine administered orally, once a day, at doses up to 1.4 mg/kg/day for approximately 6 weeks given in the morning is superior to placebo in children with ADHD

SECONDARY OUTCOMES:
Test the hypothesis that atomoxetine administered once daily in the evening provides superior efficacy compared with placebo in children with ADHD
Test the hypothesis that atomoxetine administered once daily in the morning provides superior efficacy in the evenings compared with placebo in children with ADHD
Test the hypothesis that atomoxetine administered once daily in the morning provides superior efficacy in the mornings (before daily dosing, i.e., nearly 24 hrs since last dosing) compared with placebo in children with ADHD based on the CGIP-M
To assess the effect of dosing atomoxetine in the morning versus placebo on measures of executive functioning
Test the hypothesis that atomoxetine administered once daily in the morning provides superior efficacy compared with placebo for measures of adaptive functioning in children with ADHD
Test the hypothesis that atomoxetine administered once daily in the evening provides superior efficacy in the evenings (before daily dosing, i.e., nearly 24 hrs since last dosing) compared with placebo in children with ADHD
Test the hypothesis that atomoxetine administered once daily in the morning provides superior efficacy in the mornings (before daily dosing, i.e., nearly 24 hrs since last dosing) compared with placebo in children with ADHD
To examine the onset of action during the first week of treatment in the morning versus in the evening versus placebo
To assess the effect of dosing atomoxetine in the evening versus placebo on measures of executive functioning
To compare morning versus evening dosing versus placebo as assessed by the CGI-ADHD-S
To assess the safety and tolerability of atomoxetine dosed in the morning versus in the evening versus placebo

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio, United States

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- [Derived] Newcorn JH, Sutton VK, Zhang S, Wilens T, Kratochvil C, Emslie GJ, D'souza DN, Schuh LM, Allen AJ. Characteristics of placebo responders in pediatric clinical trials of attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2009 Dec;48(12):1165-72. doi: 10.1097/CHI.0b013e3181bc730d. PMID 19858759
- [Derived] Block SL, Kelsey D, Coury D, Lewis D, Quintana H, Sutton V, Schuh K, Allen AJ, Sumner C. Once-daily atomoxetine for treating pediatric attention-deficit/hyperactivity disorder: comparison of morning and evening dosing. Clin Pediatr (Phila). 2009 Sep;48(7):723-33. doi: 10.1177/0009922809335321. Epub 2009 May 6. PMID 19420182
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com